CLINICAL TRIAL: NCT00434655
Title: Laparoscopic Adjustable Gastric Banding Versus Laparoscopic Sleeve Gastrectomy: A Prospective Trial
Brief Title: Laparoscopic Adjustable Gastric Banding Versus Laparoscopic Sleeve Gastrectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: North Texas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Esteban Varela MD,MPH, North Texas VA
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-010
Record Dates: First submitted 2007-02-09; First posted 2007-02-13 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-12

CONDITIONS: Morbid Obesity
Keywords: Morbid obesity; Bariatric surgery; Obesity surgery; Gastric banding; Sleeve gastrectomy
MeSH Terms: conditions — Obesity, Morbid

ARMS (2):
- 1 LAP BAND (Active Comparator)
  Interventions: Procedure: Laparoscopic restrictive procedure
- 2 Sleeve gastrectomy (Experimental)
  Interventions: Procedure: Laparoscopic restrictive procedure

INTERVENTIONS:
Procedure: Laparoscopic restrictive procedure — Morbidly Obese VETERANS will receive one of two laparoscopic bariatric restrictive procedures.

SUMMARY:
* The investigators aim to determine the clinical and metabolic outcomes of two available bariatric restrictive procedures: laparoscopic adjustable gastric banding (LAP-BAND) and laparoscopic sleeve gastrectomy for the treatment of morbid obesity (BMI > 35 with comorbidities or BMI > 40) in VETERANS.
* The investigators hypothesize that the short and long term outcomes between laparoscopic adjustable gastric banding (LAP-BAND) and sleeve gastrectomy are similar in VETERANS.

DETAILED DESCRIPTION:
This is a bariatric surgery Phase 3 prospective trial.

ELIGIBILITY:
Inclusion Criteria:

* Morbidly obese VETERANS ONLY (BMI>35 with comorbidities or BMI > 40)
* Age > 18 y/o

Exclusion Criteria:

* Pregnancy
* Severe uncontrolled medical or psychiatric conditions
* Previous bariatric surgery
* Multiple previous abdominal surgeries

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Short and long term clinical outcomes | 5 years

SECONDARY OUTCOMES:
Metabolic outcomes | 5 years
Esophago-gastric physiology | 2 years
Hormonal physiology | 5 years
Procedure costs | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Esteban Varela, MD, Principal Investigator — VA North Texas
Locations (1):
- VA North Texas, Dallas, Texas, United States